CLINICAL TRIAL: NCT04101383
Title: A Randomized Double Blinded Two-way Crossover Single-dose Pharmacokinetics and Pharmacodynamics Study of RinGlar® (LLC "GEROPHARM", Russia) Versus Lantus® (Sanofi-Aventis) in Type 1 Diabetes Mellitus Patients Using the Euglycemic Clamp Technique
Brief Title: A Study to Compare Pharmacokinetics and Pharmacodynamics of RinGlar® to Lantus® in Type 1 Diabetes Mellitus Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geropharm (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GLARGIN-CL
Record Dates: First submitted 2019-09-23; First posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Clamp Study
Keywords: Pharmacokinetics; Pharmacodynamics; Insulin glargine
MeSH Terms: interventions — Insulin Glargine

STUDY DESIGN:
Intervention Model Description: two-way crossover
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study was blinded for Sponsor, investigators and analytical laboratory
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RinGlar® (Experimental): Single subcutaneous administration of RinGlar® in dose 0.6 Units/kg
  Interventions: Drug: RinGlar®
- Lantus® (Active Comparator): Single subcutaneous administration of Lantus® in dose 0.6 Units/kg
  Interventions: Drug: Lantus®

INTERVENTIONS:
Drug: RinGlar® — Single subcutaneous administration of RinGlar® in dose 0.6 Units/kg
  Other Names: insulin glargine
  Arms: RinGlar®
Drug: Lantus® — Single subcutaneous administration of Lantus® in dose 0.6 Units/kg
  Other Names: insulin glargine
  Arms: Lantus®

SUMMARY:
Pharmacokinetics and pharmacodynamics study of 2 formulation of insulin glargine (RinGlar® GEROPHARM vers. Lantus® Sanofi-Aventis)

DETAILED DESCRIPTION:
A randomized double blinded two-way crossover single-dose pharmacokinetics and pharmacodynamics study of RinGlar® (LLC "GEROPHARM", Russia) versus Lantus® (Sanofi-Aventis) in Type 1 Diabetes Mellitus Patients using the euglycemic clamp technique

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent.
2. Caucasian males having confirmed diabetes mellitus type 1 (WHO criteria) for at least 12 months prior to screening.
3. Age of 18-65 (both incl.).
4. HbA1С ≤ 8,0 %.
5. Insulin therapy in stable doses at least 3 months. Total dose of insulin ≤ 1,2 IU/kg per day.
6. At least 6 months of Lantus use.
7. C-peptide ≤ 0,3 nM/L (or 0,5 ng/mL).
8. Body mass index equal to 18.5-32.0 kg/m2.
9. Subject must use, with their partner, methods of highly effective contraception throughout the study.
10. Subject is able and willing to comply with the requirements of the study protocol.

Exclusion Criteria:

1. Acute inflammatory diseases within 3 weeks before the screening period.
2. History or presence of uncontrolled diabetes mellitus for 6 months prior to screening.
3. Clinically significant diabetes mellitus complications (proliferative retinopathy, severe diabetic neuropathy, diabetic nephropathy (CKD-EPI < 60 mL/min/1,73 m2), diabetic foot).
4. Clinically significant deviations in basic vital signs (blood pressure, heart rate, respiration rate, body temperature), ECG and lab tests.
5. Deep vein thrombosis of lower extremities in a history of life or in a family history.
6. Taking medications (excl. insulin and ACE-inhibitors), phytopreparations, biologically active supplements less than 14 days before screening.
7. Donor blood donation or another blood loss, less than 3 months before the study.
8. Recovery after surgery process.
9. Mental, physical and other reasons that do not allow to adequately assess their behavior and properly fulfill the conditions of the research protocol, including psychiatric disorders.
10. History of significant drugs abuse conditions for 3 years prior to screening.
11. Positive testing for drugs.
12. Receiving more than 10 units. alcohol per week (1 unit of alcohol is equivalent to 0.5 liters of beer, 200 ml of wine or 50 ml of strong alcohol) or anamnestic information about alcoholism.
13. Positive testing for alcohol.
14. Nicotine dependence (use of tobacco less than 6 months before the start of screening).
15. Positive test results for hepatitis C or hepatitis B, HIV, syphilis.
16. Presence of suspicions of an inflammatory disease of the urinary system as a result of urinalysis.
17. Weighed allergic anamnesis.
18. Presence of oncology disease in the anamnesis 5 years prior the start of screening.
19. Organ transplantation in anamnesis (excl. cornea transplantation at least 3 month prior the IP administration).
20. Participation in a clinical trial of any medications less than 3 months before the IP administration.
21. Any other conditions that make it difficult, according to the informed opinion of the investigating physician, that volunteer participation in studies.
22. History of hypersensitivity to insulin, heparin and excipients of the drugs using in study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2017-10-16 (Actual); Primary Completion 2018-02-16 (Actual); Study Completion 2018-02-16 (Actual)

PRIMARY OUTCOMES:
AUC GIR(0-t) | 0 hours (pre-dose), as well as at, 30, 60, 90, 120, 150, 180, 210, 240, 270, 300, 330, 360, 420, 480, 540, 600, 660, 720, 780, 840, 900, 960, 1020, 1080, 1140, 1200, 1260, 1320, 1380, 1440 minutes post-dose
  Pharmacodynamic of insulin glargine by Assessment of GIR Area Under the Curve From Time Zero Extrapolated to "t" (AUC(0-t))
AUC(0-t) | -60, -30 and 0 hours (pre-dose), as well as at, 30, 60, 90, 120, 150, 180, 210, 240, 270, 300, 330, 360, 420, 480, 540, 600, 660, 720, 780, 840, 900, 960, 1020, 1080, 1140, 1200, 1260, 1320, 1380, 1440 minutes post-dose
  Pharmacokinetics of insulin glargine by Assessment of Area Under the Curve From Time Zero Extrapolated to "t" (AUC(0-t))

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Endocrinology Research Centre, Moscow
  - Almazov National Medical Research Centre, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No